CLINICAL TRIAL: NCT02861417
Title: Timed Sequential Busulfan and Post Transplant Cyclophosphamide for Allogeneic Transplantation
Brief Title: Busulfan, Fludarabine Phosphate, and Post-Transplant Cyclophosphamide in Treating Patients With Blood Cancer Undergoing Donor Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0137; NCI-2017-00614 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0137 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; High Risk Acute Myeloid Leukemia; High Risk Myelodysplastic Syndrome; Lymphoproliferative Disorder; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent High Risk Myelodysplastic Syndrome; Recurrent Hodgkin Lymphoma; Recurrent Myelodysplastic Syndrome; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoproliferative Disorders; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Busulfan; Cyclophosphamide; fludarabine; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group I (haploidentical donor transplant, chemotherapy) (Experimental): Patients receive busulfan IV over 3 hours on days -13, -12, and -6 to -3, thiotepa IV over 4 hours on day -7, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months and mycophenolate mofetil PO TID.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus; Drug: Thiotepa
- Group II (matched donor transplant, chemotherapy) (Experimental): Patients receive busulfan IV over 3 hours on days -13, -12, and -6 to -3, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tacrolimus
- Group III (haploidentical donor transplant, chemotherapy) (Experimental): Patients receiving haploidentical related donor transplant, diagnosis of myelofibrosis, > 60 years old, or patients with comorbidity scores > 3 will go in Group 3 or 4. If patients with comorbidity score > 3, then the principal investigator is the final arbiter of eligibility for comorbidity score > 3. Busulfan is administered at the dose calculated to achieve a total (including first two doses delivered on day -20 and day -13) system exposure of 20,000 +/- 12% uMol-min based on the pharmacokinetic studies.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus; Drug: Thiotepa
- Group IV (matched donor transplant, chemotherapy) (Experimental): Patients receiving haploidentical related donor transplant, diagnosis of myelofibrosis, > 60 years old, or patients with comorbidity scores > 3 will go in Group 3 or 4. If patients with comorbidity score >3, then the principal investigator is the final arbiter of eligibility for comorbidity score > 3. Busulfan is administered at the dose calculated to achieve a total (including first two doses delivered on day -20 and day -13) system exposure of 20,000 +/- 12% uMol-min based on the pharmacokinetic studies.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tacrolimus
- Group V (haploidentical donor transplant, chemotherapy) (Experimental): Patients receive busulfan IV over 3 hours on days -20, -13, and -6 to -3, a lower dose of thiotepa IV over 4 hours on day -7, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months and mycophenolate mofetil PO TID.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus; Drug: Thiotepa
- Group VI (matched or haploidentical transplant, chemotherapy) (Experimental): Patients receiving fully matched or haploidentical donor transplant receive busulfan IV over 3 hours on days -20, -13, and -6 to -3, a lower dose of thiotepa IV over 4 hours on day -7, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months and mycophenolate mofetil PO TID.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Drug: Tacrolimus; Drug: Thiotepa

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo stem cell transplantation
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
  Arms: Group I (haploidentical donor transplant, chemotherapy); Group III (haploidentical donor transplant, chemotherapy); Group V (haploidentical donor transplant, chemotherapy); Group VI (matched or haploidentical transplant, chemotherapy)
Other: Pharmacological Study — Correlative studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1'',1''''-Phosphinothioylidynetrisaziridine; Girostan; N,N'', N''''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
  Arms: Group I (haploidentical donor transplant, chemotherapy); Group III (haploidentical donor transplant, chemotherapy); Group V (haploidentical donor transplant, chemotherapy); Group VI (matched or haploidentical transplant, chemotherapy)

SUMMARY:
This phase II trial studies the side effect of busulfan, fludarabine phosphate, and post-transplant cyclophosphamide in treating patients with blood cancer undergoing donor stem cell transplant. Drugs used in chemotherapy, such as busulfan, fludarabine phosphate and cyclophosphamide work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy such as busulfan and fludarabine phosphate before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving cyclophosphamide after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety of timed sequential busulfan and fludarabine conditioning regimen and post transplant cyclophosphamide as determined by day 100 non-relapse mortality in patients undergoing allogeneic transplantation: from matched donors; from mismatched (haploidentical) donors.

SECONDARY OBJECTIVE:

I. To evaluate efficacy of this therapy and to compare outcomes between recipients of matched and mismatched donors by studying the following endpoints: graft versus host disease (GVHD)-free/relapse free survival; relapse-free survival; overall survival; non-relapse mortality; relapse rate; time to neutrophil and platelet engraftment; incidence of acute and chronic GVHD; grade 3 and 4 adverse events.

TERTIARY OBJECTIVE:

I. To study impact of timed sequential busulfan therapy and post-transplant cyclophosphamide on immune reconstitution and cytokines levels post-transplant.

OUTLINE: Patients are assigned to 1 of 4 groups.

GROUP I (FROM HAPLOIDENTICAL DONOR): Patients receive busulfan intravenously (IV) over 3 hours on days -13, -12, and -6 to -3, thiotepa IV over 4 hours on day -7, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or orally (PO) twice daily (BID) for up to 3 months and mycophenolate mofetil PO thrice daily (TID).

GROUP II (FROM MATCHED DONOR): Patients receive busulfan IV over 3 hours on days -13, -12, and -6 to -3, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months.

GROUP III and GROUP IV: Patients receiving haploidentical related donor transplant, diagnosis of myelofibrosis, > 60 years old, or patients with comorbidity scores > 3 will go in Group 3 or 4. If patients with comorbidity score > 3, then the principal investigator is the final arbiter of eligibility for comorbidity score > 3. Busulfan is administered at the dose calculated to achieve a total (including first two doses delivered on day -20 and day -13) system exposure of 20,000 +/- 12% uMol-min based on the pharmacokinetic studies.

GROUP V and GROUP VI: Patients receive busulfan IV over 3 hours on days -20, -13, and -6 to -3, a lower dose of thiotepa IV over 4 hours on day -7, fludarabine phosphate IV over 1 hour on days -6 to -3. Patients undergo stem cell transplantation IV on day 0. Patients then receive cyclophosphamide IV over 3 hours on days 3 and 4. Beginning on day 5, patients receive tacrolimus IV continuously or PO BID for up to 3 months and mycophenolate mofetil PO TID.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk hematologic malignancies with anticipated poor prognosis with non transplant therapy, including those in remission or with induction failure and after treated or untreated relapse; Diagnoses to be included a) Acute myeloid leukemia; b) Acute lymphocytic leukemia; c) Chronic myeloid leukemia; d) Chronic lymphoproliferative disorder; e) Myelodysplastic syndrome; f) Myeloproliferative syndromes; g) Non-Hodgkin's lymphoma; h) Hodgkin's Lymphoma; i) Multiple myeloma
* Patients must have a haploidentical related donor or a fully matched related or unrelated donor
* Performance score of >= 70 by Karnofsky/Lansky or performance score (PS) 0 to 1 (Eastern Cooperative Oncology Group [ECOG] =< 1)
* Left ventricular ejection fraction >= 50%
* Adequate pulmonary function with forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% of expected corrected for hemoglobin and/or volume; children unable to perform pulmonary function tests (e.g., less than 7 years old) pulse oximetry of >= 92% on room air
* Creatinine clearance (calculated creatinine clearance by Cockcroft-Gault using adjusted body weight if actual body weight is 20% greater than ideal is permitted) should be > 50 ml/min
* Bilirubin =< 2 x the upper limit of normal (except with patients high indirect bilirubin due to Gilbert's syndrome, hypersplenism, or hemolysis)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 200
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization; women of child bearing potential must be willing to use an effective contraceptive measure while on study
* Patient or patient's legal representative able to sign informed consent

Exclusion Criteria:

* Human immunodeficiency virus (HIV) seropositivity
* Uncontrolled infections
* Patients with comorbidity score > 3; the principal investigator is the final arbiter of eligibility for comorbidity score > 3
* Prior allogeneic transplant
* Patients with active hepatitis B and C
* Patients with prior coronary artery disease
* Patients who received inotuzumab and/or gemtuzumab in the past

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Non-relapse mortality rate | 100 days
  The proportion of patients with non-relapse mortality will be reported separately by arm, along with the corresponding 95% Bayesian credible interval.

SECONDARY OUTCOMES:
Graft versus host disease-free survival/relapse free survival | Up to 3 years
  Will be calculated from the time of transplant by the method of Kaplan and Meier. Patients with matched donors will be compared to patients with mismatched donors by the log-rank test. Cox proportional hazards regression analysis will be used to assess the association between these survival parameters and clinical and treatment covariates of interest.
Relapse-free survival | Up to 3 years
  Will be calculated from the time of transplant by the method of Kaplan and Meier. Patients with matched donors will be compared to patients with mismatched donors by the log-rank test. Cox proportional hazards regression analysis will be used to assess the association between these survival parameters and clinical and treatment covariates of interest.
Overall survival | Up to 3 years
  Will be calculated from the time of transplant by the method of Kaplan and Meier. Patients with matched donors will be compared to patients with mismatched donors by the log-rank test. Cox proportional hazards regression analysis will be used to assess the association between these survival parameters and clinical and treatment covariates of interest.
Non-relapse mortality | Up to 3 years
  The proportion of patients with non-relapse mortality will be reported separately by arm, along with the corresponding 95% Bayesian credible interval.
Relapse rate | Up to 3 years
  Will be observed.
Time to platelet and neutrophil engraftment | Up to 3 years
  Will be calculated from the time of transplant and estimated by the Kaplan-Meier method. Distributions will be compared between patients with matched and mismatched donors via the log-rank test.
Incidence of acute and chronic graft versus host disease | Up to 3 years
  Will be estimated using the method of Gooley, and the method of Fine and Gray will be used to model the incidence by disease and clinical characteristics of interest, including matched versus mismatched donors.
Incidence of grade 3 and 4 adverse events | Up to 3 years
  Descriptive statistics will be used to summarize adverse events by treatment arm. The number and proportion of subjects with treatment emergent adverse events will be reported and compared between patients with matched and mismatched donors by using Fisher's exact test. Frequency counts and percentages will also be presented of subjects with serious adverse events and adverse events leading to withdrawal. Graphical summaries will be used where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Uday R Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Popat UR, Pasvolsky O, Bassett R Jr, Mehta RS, Olson A, Chen J, Alousi AM, Al-Atrash G, Bashir Q, Gulbis AM, Hosing CM, Im JS, Kebriaei P, Khouri I, Marin D, Nieto Y, Oran B, Saini N, Shigle TL, Srour SA, Ramdial JL, Rezvani K, Qazilbash MH, Andersson BS, Champlin RE, Shpall EJ. Myeloablative fractionated busulfan for allogeneic stem cell transplant in older patients or patients with comorbidities. Blood Adv. 2023 Oct 24;7(20):6196-6205. doi: 10.1182/bloodadvances.2023010850. PMID 37611156
- See also: MD Anderson Cancer Center — http://www.mdanderson.org